CLINICAL TRIAL: NCT05312164
Title: Physio-Anatomy Clinical Data Collection Study
Status: Recruiting | Type: Observational
Sponsor: Gentuity, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 003785
Record Dates: First submitted 2022-03-18; First posted 2022-04-05 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Coronary Stenosis
MeSH Terms: conditions — Coronary Stenosis | interventions — Angiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Candidates for PCI: Patients undergoing diagnostic cardiac catheterization/PCI.
  Interventions: Device: HF-OCT Imaging; Device: FFR Pressure Wire; Device: Angiography

INTERVENTIONS:
Device: HF-OCT Imaging — Subjects undergo HF-OCT imaging of stenosed coronary arteries
Device: FFR Pressure Wire — Subjects undergo FFR physiology assessment of stenosed coronary arteries
Device: Angiography — Subjects undergo angiography imaging of stenosed coronary arteries

SUMMARY:
This is an on-label clinical study design intended for the collection of three different types of interventional procedural data using FDA-cleared cardiac catheterization technologies and drugs, each used according to its product labeling and standard practice of medicine.

DETAILED DESCRIPTION:
These devices and drugs are commonly used for patient evaluation during PCI procedures performed by Interventional Cardiologists. The three device technologies used in a single catheterization laboratory visit for assessment of the coronary arteries include:

* A coronary angiography imaging system to X-ray the coronary arteries for the evaluation of vessel narrowing or blocking.
* Pressure guidewire from one or more manufacturers for the measurement of coronary physiology parameters.
* Gentuity® HF-OCT Imaging System with Vis-Rx® Micro-Imaging catheter for imaging and sizing of the stenosed coronary arteries.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age.
* Patients provide written informed consent.
* Clinical presentation consistent with suspected coronary disease.
* Patients who are candidates for PCI and scheduled for coronary diagnostics in the cardiac catheter lab with the intent to perform a physiological assessment for de novo lesions with stenosis, if clinically indicated.

Exclusion Criteria:

* Presence of acute ST Elevation Myocardial Infarction (STEMI) at the time of the cath lab procedure.
* Contraindication for FFR examination or administration of vasodilators.
* Bacteremia or sepsis.
* Major coagulation system abnormalities.
* Severe hemodynamic instability or shock.
* Heart Failure NYHA Class IV.
* Severe valvular heart disease.
* Prior heart transplant.
* Acute renal failure based on diagnostic practice of the treating physician at time of screening.
* Patient is pregnant.
* Patient is currently enrolled in another clinical study that may impact the results of this study.
* Patient has other co-morbid condition(s) that, in the opinion of the Investigator, could limit their

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are candidates for PCI who already have a scheduled visit to the cardiac cath lab.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Collection of angiography images, HF-OCT images, and FFR pressure wire data | 2 years
  There are no efficacy or safety outcomes in this study. This study is a simple data collection study to help the sponsor develop next-generation HF-OCT software. Pressure wire data will be paired with HF-OCT images and angiography images for analysis to determine if the HF-OCT imaging technology can predict FFR physiology information from the OCT pullback.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Veteran's Administration Palo Alto, Palo Alto, California
  - Tampa General Hospital, Tampa, Florida
  - Atlanta VA Medical Center, Decatur, Georgia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - The Christ Hospital, Cincinnati, Ohio